CLINICAL TRIAL: NCT03711032
Title: A Phase 3, Randomized, Comparator-controlled Clinical Trial to Study the Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Bacillus Calmette-Guerin (BCG) in Participants With High-risk Non-muscle Invasive Bladder Cancer (HR NMIBC) That is Either Persistent or Recurrent Following BCG Induction or That is Naïve to BCG Treatment (KEYNOTE-676)
Brief Title: Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Bacillus Calmette-Guerin (BCG) in High-Risk Non-Muscle Invasive Bladder Cancer (HR NMIBC) (MK-3475-676/KEYNOTE-676)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-676; MK-3475-676 (Other: MSD); 194713 (Other: JAPIC-CTI); jRCT2031200390 (Registry Identifier: jRCT); 2022-501817-29-00 (Registry Identifier: EU CT); U1111-1282-1555 (Registry Identifier: UTN); 2018-001967-22 (EudraCT Number)
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: High-risk Non-muscle Invasive Bladder Cancer
Keywords: programmed cell death receptor 1 (PD-1); programmed cell death ligand 1 (PD-L1); anti-PD-1; anti-PD-L1; BCG; HR NMIBC; Patient Reported Outcome (PRO)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BCG plus Pembrolizumab: Post-induction Cohort A (Arm A-1) (Experimental): Participants receive BCG (Induction and Maintenance) in combination with 200 mg pembrolizumab administered intravenously (IV) every 3 weeks (Q3W) for 35 doses (~2 years).
  Interventions: Biological: Pembrolizumab; Biological: BCG
- BCG Monotherapy: Post-induction Cohort A (Arm A-2) (Experimental): Participants receive BCG monotherapy (Induction and Maintenance).
  Interventions: Biological: BCG
- BCG plus Pembrolizumab: BCG Naïve Cohort B-Reduced Maintenance (Arm B-1) (Experimental): Participants receive BCG (Induction and reduced Maintenance) in combination with 400 mg pembrolizumab administered IV every 6 weeks (Q6W) for 9 doses (~1 year).
  Interventions: Biological: Pembrolizumab; Biological: BCG
- BCG plus Pembrolizumab: BCG Naïve Cohort B-Full Maintenance (Arm B-2) (Experimental): Participants receive BCG (Induction and full Maintenance) in combination with 400 mg pembrolizumab administered IV Q6W for 9 doses (~1 year).
  Interventions: Biological: Pembrolizumab; Biological: BCG
- BCG Monotherapy: BCG Naïve Cohort B (Arm B-3) (Experimental): Participants receive BCG monotherapy (Induction and Maintenance).
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab IV infusion of 200 mg Q3W for BCG Post-Induction Cohort (Cohort A), or IV infusion of 400 mg Q6W for BCG Naïve Cohort (Cohort B), according to randomization
  Other Names: KEYTRUDA®; MK-3475
  Arms: BCG plus Pembrolizumab: BCG Naïve Cohort B-Full Maintenance (Arm B-2); BCG plus Pembrolizumab: BCG Naïve Cohort B-Reduced Maintenance (Arm B-1); BCG plus Pembrolizumab: Post-induction Cohort A (Arm A-1)
Biological: BCG — BCG (intravesical instillation): powder for instillation fluid for intravesical use, administered during Induction and Maintenance therapy
  Other Names: TICE® BCG; OncoTICE®

SUMMARY:
Researchers are looking for new ways to treat high-risk non muscle invasive bladder cancer (HR NMIBC). NMIBC is cancer in the tissue that lines the inside of the bladder but has not spread to the bladder muscle or outside of the bladder. High-risk means NMIBC may have a high chance of getting worse or coming back after treatment.

The goals of this study are to learn: 1. If more people who receive pembrolizumab with Bacillus Calmette-Guerin (BCG) have no signs of cancer in their body and live longer without the cancer growing, spreading, or coming back compared to people who receive BCG alone. 2. About the safety and how well people tolerate BCG alone or in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Have locally and blinded independent central review (BICR)-confirmed histological diagnosis of high-risk non-muscle invasive (T1, high grade Ta and/or CIS) UC of the bladder
* Has undergone cystoscopy/ transurethral resection of bladder tumor (TURBT) to remove all resectable disease
* Has provided tissue for biomarker analysis
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Has adequate organ function
* During the treatment period and for ≥7 days after the last dose of BCG, male participants are EITHER abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent, OR, must agree to use contraception unless confirmed to be azoospermic
* Female participants who are not pregnant, not breastfeeding, and either not a woman of child bearing potential (WOCBP); or are a WOCBP who agrees to use a contraception method that is highly effective or remains abstinent from heterosexual intercourse during the treatment period and for ≥7 days after the last dose of BCG or 120 days after the last dose of pembrolizumab, whichever comes last

BCG Post-induction Cohort (Cohort A) Only

* Has been treated with one adequate course of BCG induction therapy for the treatment of HR NMIBC
* Following adequate BCG induction therapy, must have persistent or recurrent HR NMIBC

Exclusion Criteria:

* Has a history of or concurrent locally advanced (i.e., T2, T3, T4) or metastatic UC
* Has concurrent extra-vesical (i.e, urethra, ureter, renal pelvis) non-muscle invasive urothelial carcinoma or a history of extra-vesical non-muscle invasive UC
* Has received prior therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks of start of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks of start of study treatment
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days of start of study treatment
* Has a known additional malignancy that is progressing or requires active treatment within the past 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has one or more of the following contraindications to BCG: prior BCG sepsis or systemic infection, total bladder incontinence, or an adverse experience to a previous BCG instillation that resulted in treatment discontinuation and precludes retreating with BCG
* Has an active infection or diagnosis requiring systemic antimicrobial therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has current active tuberculosis
* Has had an allogenic-tissue/solid organ transplant
* Has any contraindication(s) to IV contrast or is otherwise unable to have screening imaging with IV contrast performed

BCG Post-induction Cohort (Cohort A) Only - Has persistent T1 disease following an induction course of BCG

BCG Naïve Cohort (Cohort B) Only

- Has received any prior treatment with BCG for their NMIBC within the past 2 years prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1397 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2034-11-20 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate (CRR) by Blinded Independent Central Review (BICR) (Cohort A) | Up to ~3.5 years
  CRR is defined as the percentage of participants with carcinoma in situ (CIS) achieving a complete response (CR).
Event-Free Survival (EFS) (Cohort B) | Up to ~5 years
  EFS is defined as the time from randomization until urothelial carcinoma (UC)-defined event, or death due to any cause.

SECONDARY OUTCOMES:
EFS (Cohort A) | Up to ~5 years
  EFS is defined as the time from randomization until UC-defined event, or death due to any cause.
Recurrence-Free Survival (RFS) (Cohorts A and B) | Up to ~5 years
  RFS is defined as the time from randomization until the first occurrence of any UC recurrence, progression, or death due to any cause.
Overall Survival (OS) (Cohorts A and B) | Up to ~5 years
  OS is defined as the time from randomization to death due to any cause.
Disease Specific Survival (DSS) (Cohorts A and B) | Up to ~5 years
  DSS is defined as the time from randomization to death due to bladder cancer.
Time to Cystectomy (Cohorts A and B) | Up to ~5 years
  Time to cystectomy is defined as the time from a participant's randomization until the date of cystectomy.
12-Month EFS Rate (Cohort A) | 12 months after EFS (up to ~5 years)
  EFS is defined as the time from randomization until UC-defined event, or death due to any cause. The 12-month EFS rate is defined as the percentage of participants with EFS at 12 months.
Duration of Response (DOR) (Cohorts A and B) | Up to ~5 years
  DOR in participants with CIS is defined as the time from first documented CR until end of response or death due to any cause, whichever occurs first.
12-Month DOR Rate (Cohorts A and B) | 12 months after CR (up to ~4.5 years)
  The 12-month DOR Rate in participants with CIS is defined as the percentage of participants with a CR of at least 12 months duration.
Percentage of Participants Experiencing Adverse Events (AEs) (Cohorts A and B) | Up to ~5 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.
Percentage of Participants Discontinuing Study Drug Due to AEs (Cohorts A and B) | Up to ~5 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Combined Score (Cohorts A and B) | Baseline, time of last PRO assessment (up to ~2 years)
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall outcome. The change from baseline in Global Health Status/Quality of Life (EORTC QLQ-C30 Items 29 and 30) combined score will be presented.
Change from Baseline in EORTC-QLQ-C30 Physical Functioning (Items 1-5) Combined Score (Cohorts A and B) | Baseline, time of last PRO assessment (up to ~2 years)
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) combined score will be presented.
Change from Baseline in EORTC-QLQ-Non-muscle Invasive Bladder Cancer Module 24 (NMIBC24) Total Score (Cohorts A and B) | Baseline, time of last PRO assessment (up to ~2 years)
  The EORTC-QLQ-NMIBC24 is a 24-item questionnaire developed to supplement the EORTC QLQ-C30 in high-risk NMIBC patients. Each item is scored out of 4 total points (1=Not at All to 4=Very Much). All responses are transformed from 0 to 100, with a high score indicating more symptoms or problems. The change from baseline in EORTC-QLQ-NMIBC24 total score will be presented.
Change from Baseline in European Quality of Life (EuroQoL)-5 Dimensions, 5-level Questionnaire (EQ-5D-5L) Visual Analogue Score (VAS) (Cohorts A and B) | Baseline, time of last PRO assessment (up to ~2 years)
  The EQ-5D-5L VAS records the respondent's self-rated health on a 10 cm vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine". The change from baseline in EQ-5D-5L VAS will be presented.
Time to Deterioration (TTD) in the EORTC-QLQ-C30 Global Health Status/Quality of Life (Items 29 and 30) Combined Score (Cohorts A and B) | Time of last PRO assessment (up to ~2 years)
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall outcome. TTD in Global Health Status/Quality of Life is defined as the time from baseline to the first onset of a 10 point or greater decrease from baseline in the Global Health Status/Quality of Life (EORTC QLQ-C30 Items 29 and 30) combined score, with or without subsequent confirmation.
TTD in the EQ-5D-5L VAS (Cohorts A and B) | Time of last PRO assessment (up to ~2 years)
  The EQ-5D-5L VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine". TTD in EQ-5D-5L VAS is defined as the time from baseline to the first onset of a 7 point or greater decrease from baseline in EQ-5D-5L VAS, with or without subsequent confirmation, under a right-censoring rule.
CRR by BICR (Cohort B) | Up to ~3.5 years
  CRR is defined as the percentage of participants with CIS achieving a CR.
24-Month EFS Rate (Cohort B) | 24 months after EFS (Up to ~5 years)
  EFS is defined as the time from randomization until UC-defined event, or death due to any cause. The 24-month EFS rate is defined as the percentage of participants with EFS at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (206):
- United States (44):
  - Alaska Urological Institute dba Alaska Clinical Research Center ( Site 1083), Anchorage, Alaska
  - Mayo Clinic in Arizona - Phoenix ( Site 1094), Phoenix, Arizona
  - Arizona Urology Specialists (AUS)-Professional Park ( Site 1096), Tucson, Arizona
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 140)-Department of Urology/Institute of Uro, Los Angeles, California
  - University of California Irvine Medical Center ( Site 1061), Orange, California
  - Genesis Research LLC ( Site 1065), Torrance, California
  - Colorado Clinical Research ( Site 1100), Lakewood, Colorado
  - Urological Research Network ( Site 1106), Hialeah, Florida
  - Mayo Clinic in Florida-Urology ( Site 1097), Jacksonville, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center ( Site 1056), Miami, Florida
  - Woodlands Medical Specialists, PA ( Site 8002), Pensacola, Florida
  - Emory School of Medicine ( Site 1076), Atlanta, Georgia
  - Advanced Urology ( Site 1092), Roswell, Georgia
  - Northwestern Memorial Hospital ( Site 1101), Chicago, Illinois
  - Wichita Urology Group ( Site 1086), Wichita, Kansas
  - Ochsner LSU Health Shreveport - Regional Urology ( Site 1099), Shreveport, Louisiana
  - Henry Ford Health System ( Site 1062), Detroit, Michigan
  - Michigan Institute of Urology ( Site 1077), Troy, Michigan
  - Coastal Urology Associates ( Site 1055), Brick, New Jersey
  - Morristown Medical Center ( Site 1090), Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 1059), New Brunswick, New Jersey
  - St. Peter's Hospital Cancer Care Center ( Site 1087), Albany, New York
  - R.J. Zuckerberg Cancer Center ( Site 1080), Lake Success, New York
  - Veterans Affairs New York Harbor Healthcare System-PCF COE ( Site 1112), New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 1074), New York, New York
  - Associated Medical Professionals of NY ( Site 1078), Syracuse, New York
  - TriState Urologic Services PSC Inc. dba The Urology Group ( Site 1091), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center ( Site 1066), Cleveland, Ohio
  - Ohio State University Arthur G James Cancer Hospital & Richard J Solove Research Institute ( Site 10, Columbus, Ohio
  - OHSU Knight Cancer Institute ( Site 1075), Portland, Oregon
  - Oregon Urology Institute ( Site 1098), Springfield, Oregon
  - MidLantic Urology ( Site 1071), Bala-Cynwyd, Pennsylvania
  - Lancaster Urology ( Site 1079), Lancaster, Pennsylvania
  - University of Pennsylvania ( Site 1088), Philadelphia, Pennsylvania
  - Carolina Urologic Research Center ( Site 1085), Myrtle Beach, South Carolina
  - Urology Associates [Nashville, TN] ( Site 1072), Nashville, Tennessee
  - Urology Clinics of North Texas, PLLC ( Site 1064), Dallas, Texas
  - University Of Texas Southwestern Medical Center ( Site 1053), Dallas, Texas
  - Texas Oncology-Fort Worth Cancer Center ( Site 8003), Fort Worth, Texas
  - Houston Metro Urology ( Site 1111), Houston, Texas
  - Texas Oncology-Plano West ( Site 8001), Plano, Texas
  - Urology San Antonio Research ( Site 1108), San Antonio, Texas
  - University of Vermont Medical Center ( Site 1057), Burlington, Vermont
  - Urology of Virginia ( Site 1070), Virginia Beach, Virginia
- Australia (4):
  - GenesisCare North Shore ( Site 0010), St Leonards, New South Wales
  - Northern Cancer Institute. ( Site 0003), St Leonards, New South Wales
  - Sydney Adventist Hospital ( Site 0001), Wahroonga, New South Wales
  - Epworth Hospital ( Site 0009), Richmond, Victoria
- Austria (4):
  - Univ. Klinik f. Urologie Innsbruck ( Site 0051), Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen ( Site 0052), Linz, Upper Austria
  - Medizinische Universität Wien ( Site 0054), Vienna, Vienna
  - Universitaetsklinik Salzburg ( Site 0053), Salzburg
- Belgium (5):
  - UZA University Hospital Antwerp ( Site 0105), Edegem, Antwerpen
  - CHU UCL Namur Site de Godinne ( Site 0103), Yvoir, Namur
  - O.L.V. Ziekenhuis Aalst ( Site 0106), Aalst, Oost-Vlaanderen
  - AZ Maria Middelares Gent ( Site 0102), Ghent, Oost-Vlaanderen
  - UZ Gent ( Site 0101), Ghent, Oost-Vlaanderen
- Brazil (6):
  - Hospital São Carlos-Oncocentro Ce ( Site 1558), Fortaleza, Ceará
  - Hospital Erasto Gaertner-CEPEP - Pesquisa Clínica ( Site 1551), Curitiba, Paraná
  - Fundação Pio XII - Hospital de Câncer de Barretos-Unidade de Pesquisa Clínica ( Site 1553), Barretos, São Paulo
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO ( Site 1560), São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo ( Site 1559), São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 1554), São Paulo
- Canada (8):
  - Exdeo Clinical Research Inc. ( Site 0165), Abbotsford, British Columbia
  - Silverado Resarch Inc. ( Site 0155), Victoria, British Columbia
  - Horizon Health Network ( Site 0160), Moncton, New Brunswick
  - Princess Margaret Cancer Centre ( Site 0153), Toronto, Ontario
  - CIUSSS du Saguenay-Lac-St-Jean ( Site 0164), Chicoutimi, Quebec
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0157), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
  - CHUS - Hopital Fleurimont ( Site 0152), Sherbrooke, Quebec
- China (21):
  - Cancer Hospital Chinese Academy of Medical Science-Urinary Surgery ( Site 1766), Beijing, Beijing Municipality
  - Peking University First Hospital ( Site 1759), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Urinary Surgery ( Site 1755), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 1784), Chongqing, Chongqing Municipality
  - The First Affiliated hospital of Xiamen University-Urology ( Site 1776), Xiamen, Fujian
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE ( Site 1752), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University-Urology ( Site 1777), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University-Urology Surgery ( Site 1751), Guangzhou, Guangdong
  - ShenZhen People's Hospital ( Site 1778), Shenzhen, Guangdong
  - Harbin Medical University Cancer Hospital-urology ( Site 1772), Harbin, Heilongjiang
  - Henan Cancer Hospital-Urology ( Site 1770), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 1768), Wuhan, Hubei
  - Wuhan Union Hospital ( Site 1771), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 1763), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Urology ( S, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University-Urology ( Site 1773), Suzhou, Jiangsu
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 1764), Xi'an, Shaanxi
  - West China Hospital Sichuan University ( Site 1767), Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University ( Site 1769), Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital-Urology ( Site 1762), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Urology Surgery ( Site 1774), Wenzhou, Zhejiang
- Colombia (8):
  - Instituto de Cancerología-Oncology ( Site 1609), Medellín, Antioquia
  - Fundación Hospital San Vicente de Paúl - Rionegro - Centros Especializados o de Centros Especializad, Rionegro, Antioquia
  - Administradora Country S.A. - Clinica del Country ( Site 1607), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 1605), Bogotá, Bogota D.C.
  - Oncomedica S.A.-Oncomedica S.A ( Site 1604), Montería, Departamento de Córdoba
  - Oncologos del Occidente ( Site 1608), Pereira, Risaralda Department
  - Hemato Oncologos SA-Oncology ( Site 1601), Cali, Valle del Cauca Department
  - Clínica Imbanaco S.A.S ( Site 1611), Cali, Valle del Cauca Department
- Costa Rica (2):
  - CIMCA ( Site 1550), San José, Provincia de San José
  - Policlinico San Bosco ( Site 0600), San José
- Tampere University Hospital [Tampere Finland] ( Site 0201), Tampere, Pirkanmaa, Finland
- France (5):
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand-Urology ( Site 1355), Dijon, Bourgogne-Franche-Comté
  - Hôpital Foch-Urology department ( Site 1351), Suresnes, Hauts-de-Seine
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou ( Site 1353), Rennes, Ille-et-Vilaine
  - Hopital Claude Huriez - CHU de Lille ( Site 1360), Lille, Nord
  - HENRI MONDOR HOSPITAL ( Site 1357), Créteil, Seine-et-Marne
- Germany (5):
  - Klinikum Rechts der Isar. Technischen Universitaet Muenchen ( Site 0266), Munich, Bavaria
  - Klinikum Weiden ( Site 0259), Weiden in Der Oberpfalz, Bavaria
  - Universitaetsklinikum Wuerzburg ( Site 0265), Würzburg, Bavaria
  - Krankenhaus der Barmherzigen Brüder Trier-Abteilung für Urologie und Kinderurologie ( Site 0262), Trier, Rhineland-Palatinate
  - Universitaetsklinikum Jena ( Site 0252), Jena, Thuringia
- Greece (5):
  - Olympion General Clinic ( Site 0306), Pátrai, Achaia
  - General University Hospital of Patras ( Site 0302), Pátrai, Achaia
  - ATTIKON GENERAL UNIVERSITY HOSPITAL ( Site 0304), Chaïdári, Attica
  - Antikarkiniko Nosokomeio Thessalonikis THEAGENIO ( Site 0303), Thessaloniki, Central Macedonia
  - University Hospital of Larissa ( Site 0301), Larissa, Thessaly
- Guatemala (3):
  - INTEGRA Cancer Institute ( Site 1451), Guatemala City
  - Onco Go, S.A ( Site 1454), Guatemala City
  - Grupo Medico Angeles ( Site 1453), Guatemala City
- Hungary (4):
  - Pécsi Tudományegyetem Klinikai Központ-Urológiai Klinika ( Site 1304), Pécs, Baranya
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Urológiai Klinika ( Site 1303), Szeged, Csongrád megye
  - Semmelweis University-Urológiai Klinika ( Site 1301), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 1302), Debrecen
- Italy (12):
  - Ospedale Clinicizzato Santissima Annunziata ( Site 0361), Chieti, Abruzzo
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0353), Milan, Milano
  - Ospedale Mauriziano-SCDU ONCOLOGIA MEDICA ( Site 0366), Turin, Piedmont
  - Osp Generale Reg di Bolzano ( Site 0355), Bolzano, Trentino-Alto Adige
  - Azienda Ospedaliero Universitaria Careggi ( Site 0360), Florence, Tuscany
  - Azienda USL 8 di Arezzo-Medical Oncology ( Site 0363), Arezzo
  - Istituto Tumori Giovanni Paolo II ( Site 0357), Bari
  - Ospedale San Martino ( Site 0351), Genova
  - IRCCS Ospedale San Raffaele ( Site 0362), Milan
  - Ospedale Buccheri La Ferla Fatebenefratelli ( Site 0352), Palermo
  - Policlinico Universitario A. Gemelli ( Site 0358), Roma
  - A.O.U. di Verona - Ospedale Civile Maggiore Borgo Trento ( Site 0356), Verona
- Japan (14):
  - Hirosaki University Hospital ( Site 0407), Hirosaki, Aomori
  - Ehime University Hospital ( Site 0414), Tōon, Ehime
  - University of Tsukuba Hospital ( Site 0412), Tsukuba, Ibaraki
  - St. Marianna University Hospital ( Site 0415), Kawasaki, Kanagawa
  - Kitasato University Hospital ( Site 0403), Sagamihara, Kanagawa
  - Yokosuka Kyosai Hospital ( Site 0406), Yokosuka, Kanagawa
  - Nara Medical University Hospital ( Site 0411), Kashihara, Nara
  - Hamamatsu University Hospital ( Site 0416), Hamamatsu, Shizuoka
  - Chiba Cancer Center ( Site 0401), Chiba
  - Harasanshin Hospital ( Site 0410), Fukuoka
  - Osaka International Cancer Institute ( Site 0413), Osaka
  - Osaka Metropolitan University Hospital ( Site 0404), Osaka
  - Institute of Science Tokyo Hospital ( Site 0409), Tokyo
  - Keio University Hospital ( Site 0405), Tokyo
- University Malaya Medical Centre ( Site 1180), Kuala Lumpur, Malaysia
- Netherlands (3):
  - Maastricht University Medical Centre ( Site 0453), Maastricht, Limburg
  - Erasmus MC ( Site 0451), Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht-Medical Oncology ( Site 0455), Utrecht
- Norway (2):
  - Akershus University Hospital ( Site 0553), Lorenskog, Akershus
  - Stavanger universitetssykehus ( Site 0555), Stavanger, Rogaland
- Peru (3):
  - Hospital Nacional Guillermo Almenara Irigoyen ( Site 0601), La Victoria, Lima region
  - Oncosalud ( Site 0603), Lima, Muni Metro de Lima
  - Hospital Militar Central [Lima, Peru] ( Site 0604), Lima
- Poland (12):
  - Clinical Research Center Sp. z o.o. ( Site 0674), Poznan, Greater Poland Voivodeship
  - MICS Centrum Medyczne Torun ( Site 0679), Torun, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow ( Site 0668), Krakow, Lesser Poland Voivodeship
  - Szpital Wojewódzki im. Świętego Lukasza SP ZOZ w Tarnowie ( Site 0681), Tarnów, Lesser Poland Voivodeship
  - Uniwesytecki Szpital Kliniczny we Wroclawiu ( Site 0669), Wroclaw, Lower Silesian Voivodeship
  - Urologica Praktyka Lekarska Adam Marcheluk ( Site 0654), Siedlce, Masovian Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 0653), Warsaw, Masovian Voivodeship
  - Medical Concierge Centrum Medyczne ( Site 0676), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 0678), Przemyśl, Podkarpackie Voivodeship
  - Szpital Specjalistyczny w Koscierzynie Sp. z o.o. ( Site 0671), Kościerzyna, Pomeranian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku ( Site 0655), Słupsk, Pomeranian Voivodeship
  - LIFTMED ( Site 0652), Rybnik, Silesian Voivodeship
- Portugal (6):
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 0702), Lisbon, Lisbon District
  - Unidade Local de Saude de Braga - Hospital de Braga ( Site 0705), Braga
  - Inst. Portugues de Oncologia de Coimbra Francisco Gentil EPE ( Site 0704), Coimbra
  - Inst. Portugues de Oncologia de Lisboa Francisco Gentil EPE ( Site 0708), Lisbon
  - Hospital CUF Descobertas ( Site 0706), Lisbon
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE ( Site 0701), Porto
- Puerto Rico (2):
  - Advance Urology and Laparoscopic Center ( Site 0757), Ponce
  - Ad-Vance Medical Research ( Site 0756), Ponce
- South Korea (4):
  - Asan Medical Center ( Site 0804), Songpagu, Seoul
  - Korea University Anam Hospital ( Site 0801), Seoul
  - Seoul National University Hospital ( Site 0802), Seoul
  - Samsung Medical Center ( Site 0803), Seoul
- Spain (10):
  - Hospital Universitario Lucus Augusti ( Site 0852), Lugo, La Coruna
  - Hospital Universitario Quiron Madrid ( Site 0862), Pozuelo de Alarcón, Madrid, Comunidad de
  - Clinica Universitaria de Navarra ( Site 0863), Pamplona, Navarre
  - Fundacio Puigvert ( Site 0864), Barcelona
  - Hospital Universitario Gregorio Maranon ( Site 0854), Madrid
  - Clinica Universitaria Navarra - Madrid ( Site 0860), Madrid
  - MD Anderson Cancer Center Madrid ( Site 0859), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 0857), Madrid
  - Hospital Universitario La Paz ( Site 0866), Madrid
  - Hospital La Fe de Valencia ( Site 0855), Valencia
- Switzerland (3):
  - Universitaetsspital Basel ( Site 1201), Basel, Canton of Basel-City
  - Hopitaux Universitaires de Geneve HUG ( Site 1204), Geneva
  - Universitaetsspital Zurich ( Site 1203), Zurich
- Turkey (Türkiye) (6):
  - Ankara Universitesi Tip Fakultesi Hastanesi ( Site 0966), Ankara
  - Eskisehir Osmangazi Universitesi Hastanesi ( Site 0953), Eskişehir
  - Memorial Sisli Hastanesi-Medical Oncology ( Site 0965), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 0963), Istanbul
  - Dokuz Eylul Universitesi ( Site 0959), Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi ( Site 0961), Konya
- United Kingdom (3):
  - Raigmore Hospital ( Site 1006), Inverness, Highland
  - St Bartholomew s Hospital ( Site 1008), London, London, City of
  - St Georges University Hospitals NHS Foundation Trust. ( Site 1005), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Kamat AM, Shore N, Hahn N, Alanee S, Nishiyama H, Shariat S, Nam K, Kapadia E, Frenkl T, Steinberg G. KEYNOTE-676: Phase III study of BCG and pembrolizumab for persistent/recurrent high-risk NMIBC. Future Oncol. 2020 Apr;16(10):507-516. doi: 10.2217/fon-2019-0817. Epub 2020 Mar 12. PMID 32162533
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26322&tenant=MT_MSD_9011